CLINICAL TRIAL: NCT06947512
Title: Efficacy of the Personalization of Visual Parameters and Text-to-Speech to Improve Reading Speed, Accuracy and Comprehension in Students With Learning Disorders
Brief Title: Personalization of Visual Characters and Text-to-Speech (TTS) to Support Learning in Students With Reading Difficulties
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: IRCCS Eugenio Medea (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 996
Record Dates: First submitted 2024-03-20; First posted 2025-04-27 (Actual); Last update posted 2025-05-04 (Actual); Status verified 2025-04

CONDITIONS: Developmental Dyslexia; Reading Problem
Keywords: Developmental Dyslexia; Reading Difficulties; Personalization; Visual parameters; Auditory parameters; Fonts; Text-to-Speech (TTS)
MeSH Terms: conditions — Dyslexia

STUDY DESIGN:
Intervention Model Description: Each of the participants will be tested in two conditions: with personalized parameters and with standard parameters. Their performance in reading and writing to dictation will be compared in a single-group, within-subjects model. A post-hoc comparison will also be conducted to confirm the validity of the procedure by assessing the existence of the predicted between-groups differences in reading and writing performance.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Participant (Experimental): All participants in the study will be assessed with the Seleggo Test procedure and then tested on reading and writing to dictation in the two conditions, with personalized and with standard visual and auditory parameters for text visualization and TTS
  Interventions: Device: Seleggo Test

INTERVENTIONS:
Device: Seleggo Test — Seleggo Test is a computerized procedure to identify the personalized visual and auditory parameters facilitating reading and writing for each participant. By applying these parameters to the visualization and to the TTS software during reading of school texts, the participants are expected to be facilitated in reading and understanding the text.

SUMMARY:
Previous research has shown the importance of font type, size and spacing to facilitate text reading in dyslexia. A special automatized procedure was designed to select the most favorable parameters for both text visualization and text-to-speech (TTS) conversion to be used by students with reading difficulties. The validation of its outcomes will be carried out through a systematic comparison of the use of the personalized versus standard fonts and voices in reading and writing tests.

DETAILED DESCRIPTION:
Seleggo is a free compensatory tool for dyslexic students. It is an online platform where school textbooks are transcribed and visualized on the screen in portable format (PDF) versions, characterized by special attention to graphical features and readability, and can be listened to via TTS technology. Special functions such as karaoke modality, conceptual maps building software, summary creation, verbal and visual definition search and the possibility to record and retrieve one's own notes and sketches are also provided. Each student with Specific learning Disorder (SLD) has a personal library and can choose the parameters for text visualization to facilitate reading, modifying the display of the text, choosing font, size and spacing, as well as TTS parameters, such as speed and pitch.

The availability of many options for text visualization and TTS, however, can be advantageous only as far as the students are able to choose and use parameters that objectively facilitate their reading and comprehension. Since the analysis of the literature suggests that subjective choices may be misleading and that general recommendations may not fit the individual's needs, we decided to build an automatized, as objective as possible procedure to help the students find the combination of parameters that is most likely to facilitate them in reading and studying. This procedure, composed by an initial, gross-grained subjective procedure and followed by a thorough, systematic analysis of reading and comprehension performance, was named "Seleggo test" to match the compensatory tool it was meant to complement.

The present study aims to assess the actual advantage of personalized parameter selection through the "Seleggo Test" procedure in supporting reading compared to the use of standard parameters. The working hypothesis is that children with reading disorders would benefit from personalized text features and TTS.

The recruitment of participants will take place in schools. It is foreseen that 30 participants are recruited for each of the three groups: typically Developing children (TD), Developmental Dyslexia (DD) and Special Educational Needs (SEN) - with reading difficulties).

Additional children will be recruited form patients with DD at Scientific Institute (IRCCS) E. Medea, if necessary to reach the expected number. Children will attend the third grade of primary school to the third grade of middle school (7 to 15 years old).

ELIGIBILITY:
Inclusion Criteria (for TD group):

* age 7-15 years
* no history of reading difficulties
* attends school in Italy

Exclusion Criteria (for TD group):

* special educational needs or diagnosis of neurodevelopmental disorders

Inclusion Criteria (for DD group):

* age 7-15 years
* diagnosis of Developmental Dyslexia or Specific Reading Disorder
* Attends school in Italy

Exclusion Criteria (for DD group):

* diagnosis of Intellectual Disability

Inclusion Criteria (for SEN group):

* age 7-15 years
* reported by school to have significant difficulties in reading and writing
* Attends school in Italy (at least 6 months continued schooling and exposure to the Italian language)

Exclusion Criteria (for SEN group):

* diagnosis of Intellectual Disability

Ages: 7 Years to 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 90 (Estimated)
Dates: Start 2023-02-16 (Actual); Primary Completion 2025-11 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Reading facilitation (speed), i.e. the advantage in reading performance (speed) produced by personalized parameters as compared to standard parameters | Intervention will take place during initial assessment and will last about 1,5 hours (comparison between personalized and standard parameters during the same assessment session)
  difference between reading speed (seconds to read the text displayed by the software) with personalized and with standard visual parameters
Reading facilitation (accuracy), i.e. the advantage in reading performance (accuracy) produced by personalized parameters as compared to standard parameters | Intervention will take place during initial assessment and will last about 1,5 hours (comparison between personalized and standard parameters during the same assessment session)
  difference between reading accuracy (number of errors in reading the text displayed by the software) with personalized and with standard visual parameters
Comprehension facilitation, i.e. the advantage in auditory comprehension performance produced by personalized TTS parameters as compared to standard parameters | Intervention will take place during initial assessment and will last about 1,5 hours (comparison between personalized and standard parameters during the same assessment session)
  difference between writing accuracy (number of errors in writing a pre-defined list of nonwords) for stimuli dictated with personalized and with standard auditory parameters in the TTS device

SECONDARY OUTCOMES:
possibility to discriminate TD students' reading speed from that of students with DD and SEN | about 10 months
  difference (ANOVAs) in performance (in terms of speed, expressed in seconds per syllable) on the reading tests delivered by the software, between the three groups (TD, DD and SEN)
possibility to discriminate TD students's reading accuracy from that of students with DD and SEN | about 10 months
  difference (ANOVAs) in performance (in terms of accuracy, expressed in number of errors) on the reading tests delivered by the software, between the three groups (TD, DD and SEN)
possibility to discriminate TD students' writing accuracy from that of students with DD and SEN | about 10 months
  difference (ANOVAs) in performance (in terms of accuracy, expressed in number of errors) on the writing tests delivered by the software, between the three groups (TD, DD and SEN)
validity and reliability values for the reading speed measures collected by the software | about 10 months
  Pearson's correlations between the speed measures collected during the test and the speed measures obtained on standardized reading tests (MT test of reading speed and accuracy and Assessment Battery for Developmental Reading and Spelling Disorders).
validity and reliability values for the reading accuracy measures collected by the software | about 10 months
  Pearson's correlations between the reading accuracy measures collected during the test and the accuracy measures obtained on standardized reading tests (MT test of reading speed and accuracy and Assessment Battery for Developmental Reading and Spelling Disorders).
validity and reliability values for the writing accuracy measures collected by the software | about 10 months
  Pearson's correlations between the writing accuracy measures collected during the test and the accuracy measures obtained on standardized writing tests (Assessment Battery for Developmental Reading and Spelling Disorders).

CONTACTS AND LOCATIONS:
Locations (3):
- Italy (3):
  - IRCCS E. Medea, polo di Bosisio Parini, Bosisio Parini, LC
  - IRCCS E.Medea, polo di Conegliano, Conegliano, TV
  - Associazione La Nostra Famiglia, Treviso, TV

IPD SHARING:
Plan to Share IPD: Yes
Anonymous data will be shared through the Zenodo platform
Time Frame: From the publication of the results onwards
Access Criteria: free access, for anonymous data only

REFERENCES:
- [Background] Lorusso ML, Borasio F, Panetto P, Curioni M, Brotto G, Pons G, Carsetti A, Molteni M. Validation of a Web App Enabling Children with Dyslexia to Identify Personalized Visual and Auditory Parameters Facilitating Online Text Reading. Multimodal Technologies and Interaction. 2024; 8(1):5.